CLINICAL TRIAL: NCT02660411
Title: Impact of Inhalational Versus Intravenous Anesthesia Maintenance Methods on Long-term Survival in Elderly Patients After Cancer Surgery: a Randomized Controlled Trial
Brief Title: Impact of Anesthesia Maintenance Methods on Long-term Survival
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Collaborators: Hebei Medical University Fourth Hospital (Other); The People's Hospital of Ningxia (Other); Beijing Shijitan Hospital, Capital Medical University (Other); Guizhou Provincial People's Hospital (Other); Affiliated Hospital of Qinghai University (Other); The Third Xiangya Hospital of Central South University (Other); Cancer Hospital of Guangxi Medical University (Other); Shanxi Provincial People's Hospital (Other Government); Zhongda Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Tang-Du Hospital (Other); Tianjin Nankai Hospital (Other); Shenzhen Second People's Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor and Chairman, Department of Anesthesiology and Critical Care Medicine, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2015[869]-2; ChiCTR-IPR-15006209 (Registry Identifier: Chinese Clinical Trial Registry (www.chictr.org.cn))
Record Dates: First submitted 2016-01-07; First posted 2016-01-21 (Estimated); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Aged; Neoplasms; Surgical Procedure, Operative; Anesthesia, Inhalation; Anesthesia, Intravenous; Survival
Keywords: Sevoflurane; Propofol; Aged; Neoplasm; Surgical Procedure, Operative; Long-term survival
MeSH Terms: conditions — Neoplasms; Respiratory Aspiration | interventions — Sevoflurane; Inhalation; Propofol; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sevoflurane group (Active Comparator): Anesthesia will be induced intravenously with midazolam (0.015-0.03 mg/kg), sufentanil, propofol, and rocuronium.
  Sevoflurane will be administered by inhalation for anesthesia maintenance. The concentration of inhaled sevoflurane will be adjusted to maintain the bispectral index (BIS) value between 40 and 60. Analgesia will be supplemented with remifentanil (administered by continuous infusion), sufentanil (administered by intermittent injection/continuous infusion), or fentanyl (administered by intermittent injection).
  Towards the end of surgery, sevoflurane inhalational concentration will be decreased and fentanyl/sufentanil will be administered when necessary. Sevoflurane inhalation will be stopped at the end of surgery.
  Interventions: Drug: Sevoflurane
- Propofol group (Experimental): Anesthesia will be induced intravenously with midazolam (0.015-0.03 mg/kg), sufentanil, propofol, and rocuronium.
  Propofol will be administered by intravenous infusion for anesthesia maintenance. The infusion rate of propofol will be adjusted to maintain the BIS value between 40 and 60. Analgesia will be supplemented with remifentanil (administered by continuous infusion), sufentanil (administered by intermittent injection/continuous infusion), or fentanyl (administered by intermittent injection).
  Towards the end of surgery, propofol infusion rate will be decreased and fentanyl/sufentanil will be administered when necessary. Propofol infusion will be stopped at the end of surgery.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Sevoflurane — Sevoflurane will be administered by inhalation for anesthesia maintenance. The concentration of inhaled sevoflurane will be adjusted to maintain the BIS value between 40 and 60. Sevoflurane inhalational concentration will be decreased towards the end of surgery. Sevoflurane inhalation will be stopped at the end of surgery.
  Other Names: Sevoflurane for inhalation
  Arms: Sevoflurane group
Drug: Propofol — Propofol will be administered by intravenous infusion for anesthesia maintenance. The infusion rate of propofol will be adjusted to maintain the BIS value between 40 and 60. Propofol infusion rate will be decreased towards the end of surgery. Propofol infusion will be stopped at the end of surgery.
  Other Names: Propofol for injection
  Arms: Propofol group

SUMMARY:
Surgery is one of the major treatment methods for patients with malignant tumor. And, alone with the ageing process, more and more elderly patients undergo surgery for malignant tumor. Evidence emerges that choice of anesthetics, i.e., either inhalational or intravenous anesthetics, may influence the outcome of elderly patients undergoing cancer surgery. From the point of view of immune function after surgery and invasiveness of malignant tumor cells, propofol intravenous anesthesia may be superior to inhalational anesthesia. However, the clinical significance of these effects remains unclear. Retrospective studies indicated that use of propofol intravenous anesthesia was associated higher long-term survival rate. Prospective studies exploring the effect of anesthetic choice on long-term survival in cancer surgery patients are urgently needed.

DETAILED DESCRIPTION:
It is estimated that 234.2 million major surgical procedures are undertaken every year worldwide. Surgery is one of the major treatment methods for patients with malignant tumor. And, alone with the ageing process, more and more elderly patients undergo surgery for malignant tumor. However, evidence emerges that choice of anesthetics, i.e., either inhalational or intravenous anesthetics, may influence the outcome of elderly patients undergoing cancer surgery.

A. Effects of anesthetics on immune function after surgery

The choice of general anesthetics might influence human's immune function after surgery. An international multicenter team (NCT00418457) investigated the effects of propofol-paravertebral anesthesia vs sevoflurane-opioid anesthesia on the immune function in patients after breast cancer surgery. In a small sample size (n = 32) randomized controlled trail published in 2010, postoperative serum concentrations of interleukin (IL)-1 (protumorigenic cytokine) and matrix metalloproteinases (MMP)-3/9 (associated with cancer cell invasion and metastasis) were significantly lower (P = 0.003 and 0.011, respectively), whereas that of IL-10 (antitumorigenic cytokines) was significantly higher in the propofol group than in the sevoflurane group (P = 0.001). In another small sample size (n = 10) randomized controlled trail published in 2014, serum obtained from patients who received propofol anesthesia led to greater human donor natural killer (NK) cell cytotoxicity in vitro when compared with serum from those who received sevoflurane anesthesia. In a recent small sample size (n = 28) randomized controlled trial, the levels of NK and T helper cell infiltration in breast cancer tissue were significantly higher in patients receiving propofol anesthesia than those receiving sevoflurane anesthesia (P = 0.015 and 0.03, respectively).

Similar findings were reported in patients with other malignant tumors. In a small randomized controlled trial, 30 patients with non-small-cell lung cancer randomly received either propofol or isoflurane anesthesia. The results showed that cluster of differentiation (CD)4+CD28+ percentage (P < 0.0001) and the ratio of interferon-gamma:interleukin-4 (P = 0.001) all increased significantly with propofol but no change with isoflurane anesthesia; indicating that propofol promotes activation and differentiation of peripheral T-helper cells. In another randomized controlled trial, 60 patients undergoing surgery for tongue cancer surgery randomly received total propofol, mixed (propofol induction and sevoflurane maintenance) anesthesia or total sevoflurane anesthesia. The results showed that the percentages of CD3+, CD3+CD4+, and NK cells and the ratio of CD4+/CD8+ were significantly decreased in the two sevoflurane groups, but not in the total propofol group; suggesting that propofol has less effects on cellular immune response than sevoflurane. There are also studies that reported neutral results.

The above studies suggest that, when compared with inhalational anesthesia, propofol intravenous anesthesia may have favorable effects on the immune function in patients after cancer surgery. However, care must be taken when explaining these results: (1) the sample sizes of the available studies were small; (2) the relationship between postoperative immune function changes and long-term outcomes remains unclear.

B. Effects of anesthetics on invasiveness of malignant tumor

The effects of anesthetics on invasiveness of tumor cells were mainly tested in the experimental studies, i.e., tumor cells were incubated with anesthetics in the in vitro environment. In this aspect, propofol shows somewhat favorable effects. The results of Miao et al. showed that propofol stimulation decreased the expression of MMP-2 and -9 and subsequently decreased the invasive activity of human colon cancer cells, possibly via extracellular signal-regulated kinase 1/2 (ERK1/2) down-regulation mediated through the gamma-aminobutyric acid (GABA)-A receptor. The study of Wang et al. reported that propofol inhibited invasion and metastasis, and enhanced paclitaxel-induced apoptosis of ovarian cancer cells, possibly by suppressing the Slug expression. Ecimovic et al. also reported that propofol reduced migration in both estrogen receptor-positive and -negative breast cancer cells, possibly by suppressing the Neuroepithelial Cell Transforming Gene 1 (NET1) expression.

The reported effects of various inhalational anesthetics are conflicting. Huang et al. compared the effects of propofol and isoflurane on prostate cancer cells. The results showed that propofol, at clinical relevant concentration, inhibited the activation of hypoxia-inducible factor (HIF)-1 alpha, and partially reduced cancer cell malignant activities; whereas isoflurane raised HIF-1 alpha expression, and increased the probability of proliferation and migration. The study of Benaonana et al. reported similar results, i.e., isoflurane up-regulated the expression of HIFs, and increased the growth and malignant potential of renal cancer cells. On the other hand, sevoflurane and desflurane show opposite effects. Multiple studies found that sevoflurane inhibited the proliferation and migration, and induced apoptosis of lung cancer cells. Müller-Edenborn et al. also reported that volatile anesthetics (sevoflurane and desflurane) reduced invasion of colorectal cancer cells through down-regulation of matrix metalloproteinase-9.

So far, the clinical significance of anesthetics on the invasiveness of malignant tumors is still lacking.

C. Effect of anesthetics on long-term outcome after cancer surgery

Studies in this aspect are very limited. In the study of Enlund et al., 2838 patients who underwent breast cancer or colorectal cancer surgery were retrospectively analyzed, among them 1935 received sevoflurane anesthesia and 903 propofol anesthesia. The 1-year and 5-year survival rates were higher in propofol-anesthetized patients than in sevoflurane-anesthetized ones (differences in overall survival rate were 4.7%, P = 0.004 and 5.6%, P < 0.001, respectively). However, the differences were not statistically significant after adjusting for confounding factors. In a recent study, Wigmore et al. retrospectively investigated 11,395 patients after cancer surgery. After exclusions and propensity matching, 2,607 patients remained in each of the inhalational anesthesia group or total intravenous anesthesia group. The results showed that, after a median follow-up duration of 2.66 years (95% confidence interval [CI] 2.62-2.69), volatile inhalational anesthesia was associated with a higher risk for death after both univariate (HR 1.59, 95% CI 1.30-1.95) and multivariable analysis (HR 1.46, 95% CI 1.29-1.66).

However, in this aspect, long-term follow-up results of randomized controlled trials are still lacking. Prospective studies exploring the effect of anesthetic choice on long-term survival in cancer surgery patients are urgently needed.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be included if they meet all the following criteria:

  1. Age ≥ 65 years and < 90 years;
  2. Primary malignant tumor;
  3. Do not receive radiation therapy or chemotherapy before surgery;
  4. Scheduled to undergo surgery for the treatment of tumors, with an expected duration of 2 hours or more, under general anesthesia;
  5. Agree to participate, and give signed written informed consent.

Exclusion Criteria:

* Patients will be excluded if they meet any of the following criteria:

  1. Preoperative history of schizophrenia, epilepsy, parkinsonism or myasthenia gravis;
  2. Inability to communicate in the preoperative period (coma, profound dementia, language barrier, or end-stage disease);
  3. Critical illness (preoperative American Society of Anesthesiologists physical status classification ≥ IV), severe hepatic dysfunction (Child-Pugh class C), or severe renal dysfunction (undergoing dialysis before surgery);
  4. Neurosurgery;
  5. Other reasons that are considered unsuitable for participation by the responsible surgeons or investigators (reasons must be recorded in the case report form).

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1228 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2017-09-29 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Over survival after surgery. | Up to 5 years after surgery.
  Time from surgery to the date of all-cause death.

SECONDARY OUTCOMES:
Recurrence-free survival after surgery | Up to 5 years after surgery
  Time from surgery to the date of cancer recurrence/metastasis or all-cause death, whichever occurs first.
Event-free survival after surgery | Up to 5 years after surgery
  Time from surgery to the date of cancer recurrence/metastasis, new cancer, new serious non-cancer disease, or all-cause death, whichever occurs first.

OTHER OUTCOMES:
Quality of life in 3-year survivors after surgery. | Assessed at the end of the 3rd year after surgery.
  Quality of life is assessed with the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30).
Cognitive function in 3-year survivors after surgery. | Assessed at the end of the 3rd year after surgery.
  Cognitive function is assessed with the Telephone Interview for Cognitive Status-Modified (TICS-m).

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (17):
- China (17):
  - Department of Anesthesiology and Critical Care Medicine, Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Shijitan Hospital, Beijing, Beijing Municipality
  - Peking University Cancer Hospital, Beijing, Beijing Municipality
  - University School and Hospital of Stomatology, Beijing, Beijing Municipality
  - Cancer Hospital of Guangxi Medical University, Nanning, Guangxi
  - Shenzhen Second People's Hospital, Shenzhen, Guangzhou
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - Hebei Medical University Forth Hospital, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Zhengzhou University, Zhenzhou, Henan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Zhongda Hospital, Nanjing, Jiangsu
  - Ningxia People's Hospital, Yinchuan, Ningxia
  - Affiliated Hospital of Qinghai University, Xining, Qinghai
  - Tang-Du Hospital, Xi'an, Shaanxi
  - Shaanxi Provincial People's Hospital, Taiyuan, Shanxi
  - Shanxi Province Cancer Hospital, Taiyuan, Shanxi
  - Tianjin Nankai Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weiser TG, Regenbogen SE, Thompson KD, Haynes AB, Lipsitz SR, Berry WR, Gawande AA. An estimation of the global volume of surgery: a modelling strategy based on available data. Lancet. 2008 Jul 12;372(9633):139-144. doi: 10.1016/S0140-6736(08)60878-8. Epub 2008 Jun 24. PMID 18582931
- [Background] Deegan CA, Murray D, Doran P, Moriarty DC, Sessler DI, Mascha E, Kavanagh BP, Buggy DJ. Anesthetic technique and the cytokine and matrix metalloproteinase response to primary breast cancer surgery. Reg Anesth Pain Med. 2010 Nov-Dec;35(6):490-5. doi: 10.1097/AAP.0b013e3181ef4d05. PMID 20975461
- [Background] Buckley A, McQuaid S, Johnson P, Buggy DJ. Effect of anaesthetic technique on the natural killer cell anti-tumour activity of serum from women undergoing breast cancer surgery: a pilot study. Br J Anaesth. 2014 Jul;113 Suppl 1:i56-62. doi: 10.1093/bja/aeu200. Epub 2014 Jul 9. PMID 25009196
- [Background] Desmond F, McCormack J, Mulligan N, Stokes M, Buggy DJ. Effect of anaesthetic technique on immune cell infiltration in breast cancer: a follow-up pilot analysis of a prospective, randomised, investigator-masked study. Anticancer Res. 2015 Mar;35(3):1311-9. PMID 25750280
- [Background] Ren XF, Li WZ, Meng FY, Lin CF. Differential effects of propofol and isoflurane on the activation of T-helper cells in lung cancer patients. Anaesthesia. 2010 May;65(5):478-82. doi: 10.1111/j.1365-2044.2010.06304.x. Epub 2010 Mar 19. PMID 20337621
- [Background] Zhang T, Fan Y, Liu K, Wang Y. Effects of different general anaesthetic techniques on immune responses in patients undergoing surgery for tongue cancer. Anaesth Intensive Care. 2014 Mar;42(2):220-7. doi: 10.1177/0310057X1404200209. PMID 24580388
- [Background] Margarit SC, Vasian HN, Balla E, Vesa S, Ionescu DC. The influence of total intravenous anaesthesia and isoflurane anaesthesia on plasma interleukin-6 and interleukin-10 concentrations after colorectal surgery for cancer: a randomised controlled trial. Eur J Anaesthesiol. 2014 Dec;31(12):678-84. doi: 10.1097/EJA.0000000000000057. PMID 24614619
- [Background] Miao Y, Zhang Y, Wan H, Chen L, Wang F. GABA-receptor agonist, propofol inhibits invasion of colon carcinoma cells. Biomed Pharmacother. 2010 Nov;64(9):583-8. doi: 10.1016/j.biopha.2010.03.006. Epub 2010 May 4. PMID 20888181
- [Background] Wang P, Chen J, Mu LH, Du QH, Niu XH, Zhang MY. Propofol inhibits invasion and enhances paclitaxel- induced apoptosis in ovarian cancer cells through the suppression of the transcription factor slug. Eur Rev Med Pharmacol Sci. 2013 Jul;17(13):1722-9. PMID 23852894
- [Background] Ecimovic P, Murray D, Doran P, Buggy DJ. Propofol and bupivacaine in breast cancer cell function in vitro - role of the NET1 gene. Anticancer Res. 2014 Mar;34(3):1321-31. PMID 24596379
- [Background] Huang H, Benzonana LL, Zhao H, Watts HR, Perry NJ, Bevan C, Brown R, Ma D. Prostate cancer cell malignancy via modulation of HIF-1alpha pathway with isoflurane and propofol alone and in combination. Br J Cancer. 2014 Sep 23;111(7):1338-49. doi: 10.1038/bjc.2014.426. Epub 2014 Jul 29. PMID 25072260
- [Background] Benzonana LL, Perry NJ, Watts HR, Yang B, Perry IA, Coombes C, Takata M, Ma D. Isoflurane, a commonly used volatile anesthetic, enhances renal cancer growth and malignant potential via the hypoxia-inducible factor cellular signaling pathway in vitro. Anesthesiology. 2013 Sep;119(3):593-605. doi: 10.1097/ALN.0b013e31829e47fd. PMID 23774231
- [Background] Liang H, Gu M, Yang C, Wang H, Wen X, Zhou Q. Sevoflurane inhibits invasion and migration of lung cancer cells by inactivating the p38 MAPK signaling pathway. J Anesth. 2012 Jun;26(3):381-92. doi: 10.1007/s00540-011-1317-y. Epub 2012 Feb 17. PMID 22349744
- [Background] Wei GH, Zhang J, Liao DQ, Li Z, Yang J, Luo NF, Gu Y. The common anesthetic, sevoflurane, induces apoptosis in A549 lung alveolar epithelial cells. Mol Med Rep. 2014 Jan;9(1):197-203. doi: 10.3892/mmr.2013.1806. Epub 2013 Nov 18. PMID 24248633
- [Background] Liang H, Yang CX, Zhang B, Wang HB, Liu HZ, Lai XH, Liao MJ, Zhang T. Sevoflurane suppresses hypoxia-induced growth and metastasis of lung cancer cells via inhibiting hypoxia-inducible factor-1alpha. J Anesth. 2015 Dec;29(6):821-30. doi: 10.1007/s00540-015-2035-7. Epub 2015 May 23. PMID 26002230
- [Background] Muller-Edenborn B, Roth-Z'graggen B, Bartnicka K, Borgeat A, Hoos A, Borsig L, Beck-Schimmer B. Volatile anesthetics reduce invasion of colorectal cancer cells through down-regulation of matrix metalloproteinase-9. Anesthesiology. 2012 Aug;117(2):293-301. doi: 10.1097/ALN.0b013e3182605df1. PMID 22739763
- [Background] Enlund M, Berglund A, Andreasson K, Cicek C, Enlund A, Bergkvist L. The choice of anaesthetic--sevoflurane or propofol--and outcome from cancer surgery: a retrospective analysis. Ups J Med Sci. 2014 Aug;119(3):251-61. doi: 10.3109/03009734.2014.922649. Epub 2014 May 26. PMID 24857018
- [Background] Wigmore TJ, Mohammed K, Jhanji S. Long-term Survival for Patients Undergoing Volatile versus IV Anesthesia for Cancer Surgery: A Retrospective Analysis. Anesthesiology. 2016 Jan;124(1):69-79. doi: 10.1097/ALN.0000000000000936. PMID 26556730
- [Derived] Cao SJ, Zhang Y, Zhang YX, Zhao W, Pan LH, Sun XD, Jia Z, Ouyang W, Ye QS, Zhang FX, Guo YQ, Ai YQ, Zhao BJ, Yu JB, Liu ZH, Yin N, Li XY, Ma JH, Li HJ, Wang MR, Sessler DI, Ma D, Wang DX; First Study of Perioperative Organ Protection (SPOP1) investigators. Long-term survival in older patients given propofol or sevoflurane anaesthesia for major cancer surgery: follow-up of a multicentre randomised trial. Br J Anaesth. 2023 Aug;131(2):266-275. doi: 10.1016/j.bja.2023.01.023. Epub 2023 Jun 4. PMID 37474242
- [Derived] Zhang Y, Li HJ, Wang DX, Jia HQ, Sun XD, Pan LH, Ye QS, Ouyang W, Jia Z, Zhang FX, Guo YQ, Ai YQ, Zhao BJ, Yang XD, Zhang QG, Yin N, Tan HY, Liu ZH, Yu JB, Ma D. Impact of inhalational versus intravenous anaesthesia on early delirium and long-term survival in elderly patients after cancer surgery: study protocol of a multicentre, open-label, and randomised controlled trial. BMJ Open. 2017 Nov 28;7(11):e018607. doi: 10.1136/bmjopen-2017-018607. PMID 29187413